CLINICAL TRIAL: NCT06858475
Title: Long-term Observation Of Patient Engagement in Automated Insulin Delivery
Acronym: LOOPED
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2025/0001
Record Dates: First submitted 2025-02-21; First posted 2025-03-05 (Actual); Last update posted 2025-06-20 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 diabetes mellitus; Automated insulin delivery; Continuous glucose monitoring; Carbohydrate counting; Meal announcement
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- With device
  Interventions: Device: CONTROL-IQ (Tandem™)

INTERVENTIONS:
Device: CONTROL-IQ (Tandem™) — interaction with the CONTROL-IQ (Tandem™) hybrid closed-loop (HCL) system in individuals with type 1 diabetes

SUMMARY:
The purpose of this study is to assess the long-term evolution of patient interaction with the CONTROL-IQ (Tandem™) hybrid closed-loop (HCL) system in individuals with type 1 diabetes over 24 months. Specifically, the study examines user-initiated boluses and carbohydrate announcements to determine whether initially low-engagement users increase their involvement over time or, conversely, whether highly engaged users gradually rely more on automation.

DETAILED DESCRIPTION:
Automated insulin delivery (AID) systems have revolutionized type 1 diabetes (T1D) management, offering superior glycemic control and quality of life compared to sensor-augmented insulin pumps or multiple daily injections (MDI). However, current AID systems operate as hybrid closed-loop (HCL) systems, requiring user intervention for meal boluses, including carbohydrate counting and timely insulin administration.

Control-IQ (Tandem™) was the second AID system reimbursed by the French National Health Insurance and is now widely used in France. It combines the Tandem™ t:slim insulin pump with Dexcom™ G6 continuous glucose monitoring (CGM), adjusting basal insulin every five minutes based on glucose predictions and delivering automatic correction boluses once per hour. Despite these automation features, users must still manually initiate meal boluses, and additional correction boluses remain optional. While engagement in carbohydrate counting and timely meal announcements improves metabolic outcomes, real-world data suggest that AID benefits individuals across varying engagement levels.

Long-term data on patient behavior and engagement, particularly regarding carbohydrate announcements and the ratio of automatic to user-initiated boluses, remain limited. Understanding these patterns could reveal whether initially low-engagement users increase involvement over time or whether highly engaged users eventually rely more on automation.

This single-center, 24-month observational study will follow all T1D patients treated with Control-IQ at the Centre Hospitalier Sud-Francilien between October 2021 and October 2024.

ELIGIBILITY:
Inclusion Criteria:

* Patients using the CONTROL-IQ hybrid closed-loop system with data uploaded to the myDiabby platform at least once between October 2021 and October 2024, affiliated with the diabetology department of CHSF.

Exclusion Criteria:

* Patients with a type of diabetes other than type 1 diabetes.
* Patients who have objected to the use of their data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population will be selected from the diabetes department of a French public hospital. All eligible patients will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 453 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
number of automatic boluses | repeated measurement over 24 months (8 quarters)
  To assess the 24-month evolution of the automatic-to-user-initiated bolus ratio

SECONDARY OUTCOMES:
time spent in closed-loop mode | repeated measurement over 24 months (8 quarters)
  Measurement of the quarterly evolution, over 24 months, of the percentage of time spent in closed-loop mode (CONTROL-IQ ON)
insulin dose (UI) | repeated measurement over 24 months (8 quarters)
  Measurement of the quarterly evolution, over 24 months, of the average of total daily insulin dose (UI)
carbohydrates | repeated measurement over 24 months (8 quarters)
  Measurement of the quarterly evolution, over 24 months, of the average amount of carbohydrates reported daily in closed-loop mode (CONTROL-IQ).
glucose | Repeated measurement over 24 months (8 quarters)
  Measurement of the quarterly evolution, over 24 months, of continuous glucose monitoring parameters, including average glucose in closed-loop mode (CONTROL-IQ).
glucose management indicator | Repeated measurement over 24 months (8 quarters)
  Measurement of the quarterly evolution, over 24 months, of continuous glucose monitoring parameters, including average glucose management indicator in closed-loop mode (CONTROL-IQ).
glucose coefficient of variation | Repeated measurement over 24 months (8 quarters)
  Measurement of the quarterly evolution, over 24 months, of continuous glucose monitoring parameters, including glucose coefficient of variation in closed-loop mode (CONTROL-IQ).
percentage of time in target range (70-180 mg/dL) | Repeated measurement over 24 months (8 quarters)
  Measurement of the quarterly evolution, over 24 months, of continuous glucose monitoring parameters, including percentage of time in target range (70-180 mg/dL) in closed-loop mode (CONTROL-IQ).

CONTACTS AND LOCATIONS:
Overall Officials: Coralie AMADOU, MD, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No